CLINICAL TRIAL: NCT04328493
Title: A Multi Center Randomized Open Label Trial on the Safety and Efficacy of Chloroquine for the Treatment of Hospitalized Adults With Laboratory Confirmed SARS-CoV-2 Infection in Vietnam
Brief Title: The Vietnam Chloroquine Treatment on COVID-19
Acronym: VICO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oxford University Clinical Research Unit, Vietnam (Other)
Collaborators: Ministry of Health, Vietnam (Other Government); Hospital for Tropical Diseases, Ho Chi Minh City, Vietnam (Other); Cu Chi COVID Hospital, Vietnam (Unknown); Can Gio COVID Hospital, Vietnam (Unknown); Cho Ray Hospital (Other); National Hospital for Tropical Diseases, Hanoi, Vietnam (Other Government); Department of Health, Ho Chi Minh city (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COVID
Record Dates: First submitted 2020-03-27; First posted 2020-03-31 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: SARS-CoV-2 Infection; COVID-19
Keywords: SARS-CoV-2; COVID-19; chloroquine
MeSH Terms: conditions — COVID-19 | interventions — chloroquine diphosphate; Chloroquine

STUDY DESIGN:
Intervention Model Description: The main trial is an open label, randomised, controlled trial that will be conducted in in-patients in Ho Chi Minh City. Viet Nam. Randomization will be 1:1, stratified by study site and severity of illness, to either with or without chloroquine for 10 days. All patients will also receive a supportive care/treatment according to VN MoH's guideline for COVID-19
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (No Intervention): Patients randomized to the control arm will receive a standard of care therapy (a supportive care/treatment according to VN MoH's guideline).
- Intervention arm (Experimental): In addition to standard of care therapy, patients randomized to the intervention arm receive chloroquine phosphate as below.
  For adult ≥ 53kg: 1000mg (4 tablets) at initial dose (T=0), followed by 500mg (2 tablets) at 6 hours later (T=6), and 500mg (2 tablets) once daily for 9 days.
  For adult from 45 - 52kg: 875mg (3.5 tablets) at T=0, followed by 500mg (2 tablets) at T=6 and 500mg (2 tablets) once daily thereafter.
  For adult weighted 38 -<45 kg: 750mg (3 tablets) at T=0, followed by 375mg (1.5 tablets) at T = 6 and 375mg (1.5 tablets) once daily thereafter.
  For adult weighted <38 kg: 625mg (2.5 tablets) at T=0, followed by 375mg (1.5 tablets) at T=6 and 375mg (1.5 tablets) once daily thereafter.
  The total duration of treatment with chloroquine will be 10 days.
  Interventions: Drug: Chloroquine phosphate

INTERVENTIONS:
Drug: Chloroquine phosphate — Each chloroquine tablet contains 250mg chloroquine phosphate (or 150mg chloroquine base). Chloroquine treatment for patient is weight-based dosing.
  Chloroquine will be administered orally, as tablets. For unconscious patients chloroquine can be crushed and administered as a suspension via a nasogastric tube.
  The total duration of treatment with Chloroquine will be 10 days
  Other Names: Chloroquine
  Arms: Intervention arm

SUMMARY:
COVID-19 is a respiratory disease caused by a novel coronavirus (SARS-CoV-2) and causes substantial morbidity and mortality. There is currently no vaccine to prevent COVID-19 or therapeutic agent to treat COVID-19. This clinical trial is designed to evaluate potential therapeutics for the treatment of hospitalized COVID-19.

We hypothesis that chloroquine slows viral replication in patients with COVID-19, attenuating the infection, and resulting in more rapid declines in viral load in throat swabs. This viral attenuation should be associated with improved patient outcomes. Given the enormous experience of its use in malaria chemoprophylaxis, excellent safety and tolerability profile, and its very low cost, if proved effective then chloroquine would be a readily deployable and affordable treatment for patients with COVID-19.

The study is funded and leaded by The Ministry of Health, Vietnam.

DETAILED DESCRIPTION:
The study will start with a 10-patient prospective observational pilot study. All these patients will be subject to the same entry and exclusion criteria for the randomized trial, and undergo the same procedures. They will all receive chloroquine at the doses used in the trial (see sections below); they will not be randomized. The purpose of the pilot is to develop the study procedures for the randomized controlled trial, including the safe monitoring of patients, to refine the CRF, and to acquire some preliminary data on the safety of chloroquine in those with COVID-19.

Once the pilot study has been completed, and the data reviewed by the TSC and DMC, and the MOH ethics committee, we will then proceed to the trial. We will aim for minimum delay between completing the pilot study and starting the randomized trial.

The main study is an open label, randomised, controlled trial that will be conducted in 240 in-patients in Ho Chi Minh City. Viet Nam.

Patients will have daily assessment as per standard of care while in-patients by the hospital staff. While in-patients the study will collect the following data: peripheral oxygen saturation (pulse oximeter), respiratory rate, and FiO2. These will be recorded between 2 and 4 times per day depending on the practice of the treating site. Where recording is twice daily, one record will be made from the time period of 00:00 until 12:00, and the second recording between 12:01 and 23:59. Where the parameters are recorded four times/day they will be recorded in each of the time periods 00:00 - 06:00, 06:01 - 12:00, 12:01 - 18:00 and 18:01 - 23:59. Vitals recorded will include: FiO2, SpO2, Temp, RR HR BP. The use of ventilator or other assisted breathing device will be recorded each day.

Patients will have clinical assessment recorded as per the study schedule.

The decision to discharge patients will be at the discretion of the attending physician and depend upon the clinical status of the patient. According to current standard of care recovery and hospital discharge is dependent upon the patient having had 2 daily consecutive negative PCR throat/nose swabs. Following discharge patients will be seen on days 14, 28, 42 and 56 post-randomization.

In a subset of patients admitted to HTD we will look for ECG changes, using real-time monitoring.

Patients will have up to 1 hour ECG continuous recordings daily. The ECG recording will be downloaded from standard monitor (GE Careview) and stored electronically. ECG changes (including QT interval) will then be analyzed by machine learning.

ELIGIBILITY:
1. Laboratory-confirmed SARS-CoV-2 infection as determined by PCR, or other commercial or public health assay in any specimen < 48 hours prior to randomization, and requiring hospital admission in the opinion of the attending physician.
2. Provides written informed consent prior to initiation of any study procedures (or legally authorized representative).
3. Understands and agrees to comply with planned study procedures.
4. Agrees to the collection of OP swabs and venous blood per protocol.
5. Male or female adult ≥18 years of age at time of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-04-07 (Actual); Primary Completion 2020-09-10 (Actual); Study Completion 2020-09-10 (Actual)

PRIMARY OUTCOMES:
Viral clearance time | Up to 56 days post randomization
  Viral presence will be determined using RT-PCR to detect SARS-CoV-19 RNA. Throat/nose swabs for viral RNA will be taken daily while in hospital until there have at least 2 consecutive negative results . Virus will be defined as cleared when the patient has had ≥2 consecutive negative PCR tests. The time to viral clearance will be defined as the time following randomization to the first of the negative throat/nose swabs.

SECONDARY OUTCOMES:
Length of hospital stay | Up to 56 days post randomization
  The time since randomization to discharge between study groups
Ventilator free days | first 28 days
  The number of ventilator free days over the first 28 days of treatment
Oxygen free days | first 28 days
  The number of oxygen free days over the first 28 days of treatment
Time to death | first 7, 10, 14, 28 and 56 days since randomization
  The time to (all-cause) death following over the first 7, 10, 14, 28 and 56 days since randomization
Adverse events | Over the first 28 days (due to the prolonged half-life of Chloroquine)
  The rates of serious adverse events, rates of grade 3 or 4 adverse events
fever clearance time | Up to 56 days post randomization
  Time since randomization to the first defervescence day
Ordinal outcome scale | Up to 56 days post randomization
  WHO Ordinal outcome scale for COVID-19
Development of ARDS | Up to 56 days post randomization
  Development of ARDS defined by the Kigali criteria

CONTACTS AND LOCATIONS:
Overall Officials: Guy Thwaites, PhD. MD, Principal Investigator — University of Oxford, UK
Locations (5):
- Vietnam (5):
  - National Hospital for Tropical Diseases, Hanoi
  - Can Gio COVID Hospital, Ho Chi Minh City
  - Cho Ray Hospital, Ho Chi Minh City
  - Cu Chi COVID Hospital, Ho Chi Minh City
  - Hospital for Tropical Diseases, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Biggerstaff M, Cauchemez S, Reed C, Gambhir M, Finelli L. Estimates of the reproduction number for seasonal, pandemic, and zoonotic influenza: a systematic review of the literature. BMC Infect Dis. 2014 Sep 4;14:480. doi: 10.1186/1471-2334-14-480. PMID 25186370
- [Background] Chan JF, Kok KH, Zhu Z, Chu H, To KK, Yuan S, Yuen KY. Genomic characterization of the 2019 novel human-pathogenic coronavirus isolated from a patient with atypical pneumonia after visiting Wuhan. Emerg Microbes Infect. 2020 Jan 28;9(1):221-236. doi: 10.1080/22221751.2020.1719902. eCollection 2020. PMID 31987001
- [Background] de Wit E, Feldmann F, Cronin J, Jordan R, Okumura A, Thomas T, Scott D, Cihlar T, Feldmann H. Prophylactic and therapeutic remdesivir (GS-5734) treatment in the rhesus macaque model of MERS-CoV infection. Proc Natl Acad Sci U S A. 2020 Mar 24;117(12):6771-6776. doi: 10.1073/pnas.1922083117. Epub 2020 Feb 13. PMID 32054787
- [Background] Gao J, Tian Z, Yang X. Breakthrough: Chloroquine phosphate has shown apparent efficacy in treatment of COVID-19 associated pneumonia in clinical studies. Biosci Trends. 2020 Mar 16;14(1):72-73. doi: 10.5582/bst.2020.01047. Epub 2020 Feb 19. PMID 32074550
- [Background] Gordon CJ, Tchesnokov EP, Feng JY, Porter DP, Gotte M. The antiviral compound remdesivir potently inhibits RNA-dependent RNA polymerase from Middle East respiratory syndrome coronavirus. J Biol Chem. 2020 Apr 10;295(15):4773-4779. doi: 10.1074/jbc.AC120.013056. Epub 2020 Feb 24. PMID 32094225
- [Background] Jorge A, Ung C, Young LH, Melles RB, Choi HK. Hydroxychloroquine retinopathy - implications of research advances for rheumatology care. Nat Rev Rheumatol. 2018 Dec;14(12):693-703. doi: 10.1038/s41584-018-0111-8. PMID 30401979
- [Background] Li Q, Guan X, Wu P, Wang X, Zhou L, Tong Y, Ren R, Leung KSM, Lau EHY, Wong JY, Xing X, Xiang N, Wu Y, Li C, Chen Q, Li D, Liu T, Zhao J, Liu M, Tu W, Chen C, Jin L, Yang R, Wang Q, Zhou S, Wang R, Liu H, Luo Y, Liu Y, Shao G, Li H, Tao Z, Yang Y, Deng Z, Liu B, Ma Z, Zhang Y, Shi G, Lam TTY, Wu JT, Gao GF, Cowling BJ, Yang B, Leung GM, Feng Z. Early Transmission Dynamics in Wuhan, China, of Novel Coronavirus-Infected Pneumonia. N Engl J Med. 2020 Mar 26;382(13):1199-1207. doi: 10.1056/NEJMoa2001316. Epub 2020 Jan 29. PMID 31995857
- [Background] Liu M, He P, Liu HG, Wang XJ, Li FJ, Chen S, Lin J, Chen P, Liu JH, Li CH. [Clinical characteristics of 30 medical workers infected with new coronavirus pneumonia]. Zhonghua Jie He He Hu Xi Za Zhi. 2020 Mar 12;43(3):209-214. doi: 10.3760/cma.j.issn.1001-0939.2020.03.014. Chinese. PMID 32164090
- [Background] McChesney EW, Banks WF Jr, Fabian RJ. Tissue distribution of chloroquine, hydroxychloroquine, and desethylchloroquine in the rat. Toxicol Appl Pharmacol. 1967 May;10(3):501-13. doi: 10.1016/0041-008x(67)90089-0. No abstract available. PMID 6059665
- [Background] multicenter collaboration group of Department of Science and Technology of Guangdong Province and Health Commission of Guangdong Province for chloroquine in the treatment of novel coronavirus pneumonia. [Expert consensus on chloroquine phosphate for the treatment of novel coronavirus pneumonia]. Zhonghua Jie He He Hu Xi Za Zhi. 2020 Mar 12;43(3):185-188. doi: 10.3760/cma.j.issn.1001-0939.2020.03.009. Chinese. PMID 32164085
- [Background] Shaw K. The 2003 SARS outbreak and its impact on infection control practices. Public Health. 2006 Jan;120(1):8-14. doi: 10.1016/j.puhe.2005.10.002. Epub 2005 Nov 16. PMID 16297415
- [Background] Villegas L, McGready R, Htway M, Paw MK, Pimanpanarak M, Arunjerdja R, Viladpai-Nguen SJ, Greenwood B, White NJ, Nosten F. Chloroquine prophylaxis against vivax malaria in pregnancy: a randomized, double-blind, placebo-controlled trial. Trop Med Int Health. 2007 Feb;12(2):209-18. doi: 10.1111/j.1365-3156.2006.01778.x. PMID 17300627
- [Background] Vincent MJ, Bergeron E, Benjannet S, Erickson BR, Rollin PE, Ksiazek TG, Seidah NG, Nichol ST. Chloroquine is a potent inhibitor of SARS coronavirus infection and spread. Virol J. 2005 Aug 22;2:69. doi: 10.1186/1743-422X-2-69. PMID 16115318
- [Background] Wang M, Cao R, Zhang L, Yang X, Liu J, Xu M, Shi Z, Hu Z, Zhong W, Xiao G. Remdesivir and chloroquine effectively inhibit the recently emerged novel coronavirus (2019-nCoV) in vitro. Cell Res. 2020 Mar;30(3):269-271. doi: 10.1038/s41422-020-0282-0. Epub 2020 Feb 4. No abstract available. PMID 32020029
- [Background] White NJ, Miller KD, Churchill FC, Berry C, Brown J, Williams SB, Greenwood BM. Chloroquine treatment of severe malaria in children. Pharmacokinetics, toxicity, and new dosage recommendations. N Engl J Med. 1988 Dec 8;319(23):1493-500. doi: 10.1056/NEJM198812083192301. PMID 3054558
- [Background] Zaki AM, van Boheemen S, Bestebroer TM, Osterhaus AD, Fouchier RA. Isolation of a novel coronavirus from a man with pneumonia in Saudi Arabia. N Engl J Med. 2012 Nov 8;367(19):1814-20. doi: 10.1056/NEJMoa1211721. Epub 2012 Oct 17. PMID 23075143
- [Background] Zhao S, Lin Q, Ran J, Musa SS, Yang G, Wang W, Lou Y, Gao D, Yang L, He D, Wang MH. Preliminary estimation of the basic reproduction number of novel coronavirus (2019-nCoV) in China, from 2019 to 2020: A data-driven analysis in the early phase of the outbreak. Int J Infect Dis. 2020 Mar;92:214-217. doi: 10.1016/j.ijid.2020.01.050. Epub 2020 Jan 30. PMID 32007643
- [Background] Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, Zhao X, Huang B, Shi W, Lu R, Niu P, Zhan F, Ma X, Wang D, Xu W, Wu G, Gao GF, Tan W; China Novel Coronavirus Investigating and Research Team. A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020 Feb 20;382(8):727-733. doi: 10.1056/NEJMoa2001017. Epub 2020 Jan 24. PMID 31978945
- [Derived] Kestelyn E, Dung NTP, Lam Minh Y, Hung LM, Quan NM, Dung NT, Minh NNQ, Xuan TC, Phong NT, Ninh Thi Thanh V, Donovan J, Tu TNH, Nhat LTH, Truong NT, Man DNH, Thao HP, Ngoc NM, Lam VT, Phat HH, Phuong PM, Geskus RB, Ha VTN, Quang NN, Tran Tinh H, Tan LV, Thwaites GE, Day JN, Chau NVV; OUCRU COVID-19 Research Group. A multi centre randomized open label trial of chloroquine for the treatment of adults with SARS-CoV-2 infection in Vietnam. Wellcome Open Res. 2020 Jun 12;5:141. doi: 10.12688/wellcomeopenres.15936.1. eCollection 2020. PMID 33110944
- See also: in press — https://doi.org/10.1016/j.ijantimicag.2020.105949
- See also: World Health Organization Model List of Essential Medicines — https://apps.who.int/iris/bitstream/handle/10665/325771/WHO-MVP-EMP-IAU-2019.06-eng.pdf?ua=1
- See also: COVID-19 Coronavirus Pandemic updates — https://www.worldometers.info/coronavirus/